CLINICAL TRIAL: NCT05390086
Title: Further Development and Assessment of Tools to Measure Risk Factors for and Treatment of Thiamine Deficiency Disorders: a Comparison of Rural and Urban Contexts in Lao PDR
Brief Title: Further Development and Assessment of Tools to Measure Risk Factors for and Treatment of Thiamine Deficiency Disorders
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: Lao Tropical and Public Health Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1867468
Record Dates: First submitted 2022-05-16; First posted 2022-05-25 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Thiamine Deficiency
MeSH Terms: conditions — Thiamine Deficiency | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Standard of care — The study is being implemented among children who are seeking care at collaborating hospitals for signs and symptoms suggestive of TDD. All children will be treated by the hospital physicians following the usual hospital procedures. The study will not interfere in any with the administration of required treatments and interventions.

SUMMARY:
Thiamine deficiency, including the most severe form infantile beriberi, is a public health concern across South and Southeast Asia, where monotonous diets rely on thiamine-poor white rice. Food insecurity, food preparation and cooking practices, anti-thiamine compound consumption and culturally determined postpartum food restrictions precipitate thiamine deficiency in these high-risk regions. The risk of thiamine deficiency is highest in the first year of life, especially among exclusively or predominantly breastfed infants of mothers who are thiamine deficient themselves, as thiamine content of breastmilk is related to maternal thiamine status.

However, diagnosis of infantile thiamine deficiency is challenging due to the highly variable, non-specific clinical manifestations, referred to as thiamine deficiency disorders (TDD), that often overlap with other conditions, resulting in misdiagnosis and missed treatment opportunities, which can be fatal or have irreversible consequences. Considering that breastfed infants are at highest risk, a large proportion of infant deaths could be avoided if: 1) infants with TDD were immediately treated with thiamine when medically indicated and, importantly; 2) thiamine deficiency was prevented by improving thiamine status among breastfeeding women. The latter is important given emerging evidence of long-term neurocognitive deficits of severe and even subclinical thiamine deficiency.

In light of these diagnostic uncertainties, it was recognised that a case definition for thiamine responsive disorders (TRD) would help to better identify infants with TDD who would benefit from timely thiamine treatment. This study will test the usefulness of a recently developed case definition for TRD and practical tool in different contexts in Lao PDR where TDD have been reported. Secondly, data on diet, maternal and household risk factors for TDD in different contexts will be used to propose a community risk factor screening tool to better identify populations at risk of thiamine deficiency and help advocate for and guide planning of preventive programmes.

DETAILED DESCRIPTION:
The study's primary objective is to determine the usefulness of a TRD case definition and practical tool in identifying infants and young children that would benefit from thiamine treatment in different contexts in Lao PDR, specifically urban Vientiane and rural Luang Prabang. Clinical observers based at the participating hospitals within each country/region will record the presenting signs and symptoms of all children within the target age range (21 days - <18 months) over a one month period. For children who meet the eligibility criteria and informed consent is obtained, information will be collected on duration of hospital stay, received medical treatments, final physician diagnosis and risk factor questionnaires (see below). This data will be used to determine the sensitivity and specificity of the practical TRD case definition tool to accurately identify children who would benefit from thiamine treatment and reduce treatment uncertainties

The secondary objective is to explore risk factors associated with TDD/TRD among infants and young children and their mothers. This will help to identify potential metrics that could be included in a community risk factor screening tool to identify population groups at risk of thiamine deficiency so appropriate preventive interventions can be implemented. Data will be collected on diet and household risk factors for thiamine deficiency, including infant and young child feeding practices, maternal dietary practices, maternal health status and household socioeconomic status and food security.

ELIGIBILITY:
Inclusion Criteria:

* Infants and young children aged 21 days - <18 months presenting to the collaborating hospitals and presenting with at least one of the following signs and symptoms consistent with TDD:

  * Enlarged liver (liver edge >2 cm below the right costal margin)
  * Edema
  * Tachypnea (respiratory rate >60/min for 3-8 weeks; >50/min for 2-11 months; >40/min for 12-18 months)
  * Tachycardia (heart rate >160/min for <12 months; >120/min for 12-18 months)
  * Oxygen saturation <92%
  * Difficulty breathing (chest indrawing or nasal flaring)
  * Refusal to breastfeed or of infant formula or food for >24 hours
  * Repetitive or recurrent vomiting with no obvious other cause (>3 times in past 24 hours)
  * Persistent crying not relieved by soothing or feeding with no obvious other cause
  * Hoarse voice/cry or loss of voice
  * Nystagmus or other unusual eye movements
  * Muscle twitching
  * Loss of consciousness
  * Convulsion
  * Opisthotonos/abnormal posturing
  * Acute/flaccid paralysis

Exclusion Criteria:

* Infants and young children who do not meet any of the TDD-like signs and symptoms will not be eligible for study participation.

Ages: 21 Days to 18 Months | Sex: All
Age Groups: Child
Study Population: Infants and young children in the target age range (21 days - <18 months) who are admitted to the collaborating hospitals with at least one of the signs/symptoms suggestive of TDD will be eligible for participation.
  Mothers of all participating children will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Thiamine responsive disorder (TRD) | From hospital admission to hospital discharge
  Presenting signs and symptoms compatible with the thiamine responsive disorders (TRD) case definition and physician diagnosis of beriberi

SECONDARY OUTCOMES:
Risk factors for TDD/TRD | Baseline
  Risk factors related to TDD, TRD and physician diagnosed beriberi

CONTACTS AND LOCATIONS:
Locations (2):
- Laos (2):
  - Lao Friends Hospital for Children, Luang Prabang
  - Children's Hospital, Vientiane

IPD SHARING:
Plan to Share IPD: Yes
The complete de-identified dataset will be made publicly available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 2 years of completion of the data collection